CLINICAL TRIAL: NCT06048328
Title: Pilot of a Peer Advocacy Training Intervention to Reduce Unmet Need for Contraception in Uganda
Brief Title: Game Changers for Family Planning Peer Advocacy Program
Acronym: GC-FP
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: RAND (Other)
Collaborators: Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024-GC-FP
Record Dates: First submitted 2023-09-08; First posted 2023-09-21 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Family Planning
Keywords: contraception
MeSH Terms: interventions — Family Planning Services

STUDY DESIGN:
Intervention Model Description: parallel randomized controlled trial, with individual randomization to receive the intervention or wait-list control
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): peer-led, multi-session advocacy training group intervention
  Interventions: Behavioral: Game Changers for Family Planning
- Wait-list control (No Intervention): Usual care/no intervention

INTERVENTIONS:
Behavioral: Game Changers for Family Planning — Game Changers for Family Planning (GC-FP) intervention. The intervention will consist of 6 group sessions. The sessions will focus on stigma reduction, disclosure decision making, knowledge, and building skills for advocacy. The 2-hour, weekly sessions will be facilitated by 2 trained peers who are MC users, and conducted in Luganda using a structured manual, and group format to facilitate: sharing of experiences to build support, modeling and motivation; group problem solving and role playing to build skills and self-efficacy; and homework between sessions to practice skills and generate experiences to be processed in the group.
  Arms: Intervention

SUMMARY:
This study will adapt the Game Changers peer advocacy training model for family planning context and pilot test the feasibility, acceptability and preliminary efficacy of the intervention to empower female contraception users to advocate for contraception use among women in their social networks who have unmet need for contraception.

DETAILED DESCRIPTION:
The investigators will conduct a pilot RCT of Game Changers for Family Planning (GC-FP) with 40 female modern contraceptive (MC) users (index participants) at one rural public clinic, with 20 randomly assigned to receive the intervention (in 2 groups of 10) and 20 to the wait-list control; enrollment and randomization will be stratified by age and relationship status. Each index will recruit up to 3 social network members (alters) with unmet need for MC (max. total=120). Data will be collected at baseline and month 6 from all participants; primary outcome is alter MC use at month 6.

ELIGIBILITY:
Index participants:

Inclusion Criteria:

* MC user for past year

Social network member participant:

Inclusion Criteria:

* Not using MC, but reports trying to prevent pregnancy
* Know about the MC use of their referring index participant

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 192 (Estimated)
Dates: Start 2027-11-15 (Estimated); Primary Completion 2030-11-01 (Estimated); Study Completion 2031-07-01 (Estimated)

PRIMARY OUTCOMES:
Rate of use of modern contraceptives (social network participants) | 6 months
  Proportion of participants who use a modern contraceptive, abstracted from medical chart

SECONDARY OUTCOMES:
Mean level of engagement in family planning advocacy (index participants) | 6 months
  Mean item score on self-report scale measuring engagement in family planning advocacy

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Wagner, Principal Investigator — RAND

IPD SHARING:
Plan to Share IPD: Yes
The investigators will create public use data files that include a deidentified quantitative dataset that includes longitudinal participant-level survey scales and social network assessment data (related to the primary research questions around family planning, and moderators and mediators of the associations between the intervention and contraception use); and an excel spreadsheet with the qualitative codebook with representative quotes on key themes by subgroup, linked to ID. Only predictors and outcomes data (e.g., contraception use) will be shared; additional variables (e.g., socio-demographic characteristics) will not be included to prevent the potential and unintentional de-identification of participants.
Supporting Information: Study Protocol, SAP
Time Frame: one year after completion of study, for 12 months